CLINICAL TRIAL: NCT05233501
Title: The Effect of Low-level Laser Therapy on Levels of Tissue Plasminogen Activator and Plasminogen Activator Inhibitor 1 in Gingival Crevicular Fluid of Stage 3-4, Grade C Periodontitis Patients Received Non-surgical Periodontal Treatment.
Brief Title: Low-level Laser Therapy as an Adjunct to Non-surgical Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Ferda Pamuk Özer, Associate professor, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: interventional
Record Dates: First submitted 2022-01-13; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Periodontal Diseases; Periodontal Attachment Loss; Periodontal Disease, AVDC Stage 3; Periodontal Inflammation; Periodontal Disease, AVDC Stage 4
Keywords: periodontitis; lasers; prospective; plasminogen activator inhibitor 1; tissue plasminogen activator; low-level laser therapy; periodontal treatment
MeSH Terms: conditions — Periodontal Diseases; Periodontal Attachment Loss; Periodontitis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: a split-mouth randomized controlled clinical study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-surgical perıodontal treatment (Sham Comparator)
  Interventions: Procedure: non-surgical periodontal treatment
- non-surgical treatment+ low level laser therapy (Experimental)
  Interventions: Procedure: low level laser therapy; Procedure: non-surgical periodontal treatment

INTERVENTIONS:
Procedure: low level laser therapy — adjunctive application of low level laser therapy to non-surgical periodontal treatment
  Arms: non-surgical treatment+ low level laser therapy
Procedure: non-surgical periodontal treatment — standart periodontal therapy

SUMMARY:
The present study aimed to investigate the effects of low-level laser therapy (LLLT) as an adjunct to non-surgical periodontal treatment (NSPT) on the plasminogen-activating system in Stage 3-4, Grade C periodontitis patients.

DETAILED DESCRIPTION:
Limited data is available regarding the effects of various periodontal treatment protocols on GCF t-PA and PAI-1 levels, and the extent to which LLLT in conjunction with NSPT affects these levels in patients with Stage 3-4, Grade C periodontitis is unknown. Therefore, this study measured standard clinical outcomes and GCF t-PA and PAI-1 levels in patients with Stage 3-4 Grade, C periodontitis in order to assess the use of LLLT as an adjunct to standard NSPT.

This split-mouth study was conducted with 15 Stage 3-4, Grade C periodontitis patients and 15 healthy individuals matched for age and sex. Participants were grouped as follows: Periodontitis/NSPT (Sham); Periodontitis/NSPT+LLLT (LLLT); Periodontally Healthy (Control). LLLT was applied following NSPT and again on post-treatment Days 2 and 7. Clinical parameters were recorded at baseline (i.e. before NSPT) and on Day 30. Gingival crevicular fluid (GCF) samples were collected at baseline and during follow-up visits on Days 7, 14 and 30. GCF t-PA and PAI-1 levels were measured with ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Stage 3-4, Grade C periodontitis (at least one site with probing depth (PD) and clinical attachment level (CAL) ≥5 mm in their incisors and/or first molars and at least 6 other teeth with similar PD and CAL measurements, with alveolar bone loss confirmed by radiography; familial aggregation;
* presence of ≥16 teeth;
* no periodontal treatment in the 6 months prior to data collection;
* non-smoker

Exclusion Criteria:

* systemic problems, including a medical history of cancer, rheumatoid arthritis, diabetes mellitus, or cardiovascular disease;
* compromised immune system;
* pregnancy, menopause, or lactation;
* ongoing drug therapy that might affect the clinical characteristics of periodontitis;
* use of systemic antimicrobials during the 6 weeks prior to data collection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
the change in GCF tissue plasminogen activator | baseline and during follow-up visits on Days 7, 14 and 30.
  Gingival crevicular fluid (GCF) samples were collected before SRP treatment and on days 7, 14 and 30 of follow- up and the change of the related mediator at those time points. The Amount of the related mediator were evaluated using enzyme- linked immunosorbent assay [ELISA] kit.
  Total amounts (pg/30 s) of the mediator collected from each sample in a 30- second period were calculated and recorded for analysis.
the change in GCF plasminogen activator inhibitor 1 | baseline and during follow-up visits on Days 7, 14 and 30.
  Gingival crevicular fluid (GCF) samples were collected before SRP treatment and on days 7, 14 and 30 of follow- up and the change of the related mediator at those time points. The Amount of the related mediator were evaluated using enzyme- linked immunosorbent assay [ELISA] kit.
  Total amounts (pg/30 s) of the mediator collected from each sample in a 30- second period were calculated and recorded for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ferda Pamuk Özer, Principal Investigator — Beykent University
Locations (1):
- Beykent University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Pamuk F, Lutfioglu M, Paksoy T, Koyuncuoglu CZ, Polat NG, Cifcibasi E, Yildirim S, Kantarci A. Impact of low-level laser therapy as an adjunct to non-surgical periodontal treatment on the levels of tissue plasminogen activator and plasminogen activator inhibitor 1 in Stage 3-4, Grade C periodontitis patients: a split-mouth, randomized control study. Clin Oral Investig. 2023 Nov;27(11):6439-6449. doi: 10.1007/s00784-023-05248-z. Epub 2023 Sep 15. PMID 37709984